CLINICAL TRIAL: NCT01544413
Title: Quality Control Study for Multicenter Phase III Trial of Laparoscopic Sentinel Node Biopsy and Stomach Preserving Surgery in Early Gastric Cancer
Brief Title: Quality Control Study of Laparoscopic Sentinel Node Biopsy in Early Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Keun Won Ryu, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENORITA-2012
Record Dates: First submitted 2012-02-16; First posted 2012-03-05 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Early Gastric Cancer
Keywords: laparoscopic sentinel lymph node biopsy; quality control study; early gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic sentinel lymph node biopsy (Experimental): This is a single armed study. After endoscopic marking using Tc99m HSA and indocyanine green fluid, Laparoscopic sentinel lymph node biopsy was performed and evalute at backtable.
  Interventions: Procedure: Laparoscopic sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Laparoscopic sentinel lymph node biopsy — During the operation, endoscopic marking was perfomed using Tc 99m HSA and indocyanine green around tumor. Then we identify the sentinel lymph node with laparoscopic probe. Laparoscopic sentinel lymph nodes were dissedted and evaluated them at the backtable in the operating room.
  Other Names: Tc 99m HSA (Frosstimage); indocyanine green (IC-GREEN™ (Akorn)); laparoscopic probe (neoprobe® GDS gamma detection system)

SUMMARY:
Laparoscopic sentinel lymph node biopsy and stomach preserving surgery in ealry gastric cancer is less invasive method which can increase quality of life. Multicenter phase III trial is requred to validate this method. In this study all items which are necessary for laparoscopic sentinel lymph node biopsy are identified according to checklist and evaluated the performance completement.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma in preoperative endoscopic biopsy
* clinical stage T1-2N0
* long diameter of tumor <4cm
* distance between tumor and pylorus or cardia >2cm
* age: 20-80
* ECOG: 1 or 0
* patients will undergo laparoscopic gastrectomy

Exclusion Criteria:

* definite criteria of endoscopic submucosal dissection (size<2cm, differentiated type, no ulcer)
* no indication for surgery for cardiovascular, pulmonary disease
* pregancy
* drug allergy or previous abdominal surgery, radiotherpy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Completement of performance of laparoscopic sentinel lymph node biopsy | within 24 hours after operation
  Investigators will make out a checklist after operation for evaluating the completement of performance of laparoscopic sentinel lymph node biopsy. The checklist will be made out within 24 hours.

SECONDARY OUTCOMES:
Detection rate of laparoscopic sentinel lymph node, learning curve | upto 2 years
  Detection rate of laparoscopic sentinel lymph node is evaluated within 7 days after operation by pathological examination. Learning curve can be drawn after all cases' data are collected, so it takes upto 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Keun Won Ryu, Doctor, Principal Investigator — National Cancer Center, Korea
Locations (15):
- South Korea (15):
  - Chonnam National University Hwasun Hospital, Hwasun, Chonnam
  - National Cancer Center, Korea, Goyang-si, Gyeonggi-do
  - Ajou University School of Medicine, Suwon, Gyeonggi-do
  - Gyeongsang National University, Jinju, Gyeongsangnam-do
  - Korea University Guro Hospital, Seoul, Seoul
  - Yonsei Univeristy College of Medicine, Seoul, Seoul
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Dong-A University College of Medicine, Busan
  - Dongnam Institute of Radiological and Medical Science, Busan
  - Keimyung University School of Medicine, Daegu
  - Korea University College of Medicine, Seoul
  - Kyung Hee University Gangdong Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul